CLINICAL TRIAL: NCT06523413
Title: Effectiveness of Game Activity and Stress Ball on Preoperative Anxiety and Vital Signs
Brief Title: Effect of Game Activity and Stress Ball on Anxiety and Vital Signs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Filiz Salman Saraç, Research Assistant Dr., Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SuleymanDU_SALMAN-F-002
Record Dates: First submitted 2024-07-02; First posted 2024-07-26 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Anxiety; Arthroplasty Complications
Keywords: anxiety; vital signs; artroplasty
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group 1 (Experimental): The game designated for the group game activity will be played with the patient, the patient's relative, and the researcher before the surgery. Data will be collected by another researcher before the game is played, and measurements will be taken again using data collection tools after the group game activity.
  Interventions: Behavioral: Game activity
- Intervention Group 2 (Experimental): Patients will use the stress ball for 15 minutes before surgery. Data will be collected with data collection tools before and after using the stress ball.
  Interventions: Device: Stres Ball
- Control Group (No Intervention): No intervention will be performed on patients. Data will be collected twice before surgery.

INTERVENTIONS:
Behavioral: Game activity — A game determined by the researcher will be played with the patients in the patient room.
  Arms: Intervention Group 1
Device: Stres Ball — Patients will use the stress ball for 15 minutes.
  Arms: Intervention Group 2

SUMMARY:
This randomized controlled trial aims to determine the effect of game activity and stress ball use on preoperative anxiety and vital signs in patients undergoing total knee arthroplasty. The primary purpose of the study is to evaluate the effect of these methods (game activity, stress ball use) on patients' anxiety and vital signs. The research involves three groups: one group will engage in a game activity, another group will use a stress ball, and the control group will receive no intervention. Patients over 18 years of age who pass the Mini-Cog test, demonstrate cognitive competence and meet other sampling criteria will be included in the study. Data will be collected using the State Anxiety Scale, a vital signs and pain level form, and a descriptive characteristics form.

DETAILED DESCRIPTION:
Preoperative anxiety causes various physiological and psychological reactions. In addition, it is known that preoperative anxiety negatively affects the patient's satisfaction with the surgery, the surgical success rate, and the development of postoperative complications. Total knee arthroplasty (TKA) is a surgical procedure frequently performed today to relieve pain and restore knee joint function. Approximately 30% of patients undergoing TKA experience psychological distress before surgery. Anxiety is a problem that needs to be managed in TKA patients because it negatively affects them in the postoperative period.

Interventions such as music, funny videos, massage, meditation, hypnosis, VR glasses, and motivational interviewing have been used to reduce preoperative anxiety in adults. These methods can be applied by nurses, are low cost, and have few side effects. Gaming activities are also one of the methods used to distract patients and reduce their anxiety levels in the preoperative period. The literature shows that game-based approaches in the management of preoperative anxiety are frequently used with pediatric patients. A stress ball is a method used to draw a person's attention in a different direction by squeezing and loosening the ball held in the palm. Although the use of stress balls has not been widely studied in preoperative anxiety management, research shows that stress balls may be useful in anxiety management. Game activity and stress ball use are methods that are easy to implement and will not burden patients in terms of cost.

ELIGIBILITY:
Inclusion Criteria:

Being over 18 years old Undergoing total knee arthroplasty Having passed the Mini-Cog test Ability to understand, read, and write Turkish No hearing or speech problems Having a person accompanying the patient

Exclusion Criteria:

Not wanting to participate in the research Unstable general condition Sudden change in vital signs Having a psychological disorder and using antidepressant medication Having any psychiatric or cognitive/mental disease (e.g., dementia) Use of psychiatric medication for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Inventory (STAI-I) | The first measurement will be collected at the first encounter with the patient, the last measurements will be collected 15 minutes after the intervention in patients who underwent intervention and 1 hour after the first measurement in the control group.
  State-Trait Anxiety Inventory (STAI), developed by Spielberger (1970), is a self-assessment questionnaire consisting of short statements created to determine the level of anxiety. The scale consists of 20 items. Answers range from 1-4. The total score obtained from the scale is between 20-80. A high score indicates a high level of anxiety
Pain Level | The first measurement will be collected at the first encounter with the patient, the last measurements will be collected 15 minutes after the intervention in patients who underwent intervention and 1 hour after the first measurement in the control group.
  The intensity of the pain will be quantified using the Visual Analogue Scale (VAS). The scale is evaluated by assigning a score between 0 and 10. On the scale, the absence of pain is indicated by a rating of 0 points, while the most severe pain imaginable is indicated by a rating of 10 points.
Temperature | The first measurement will be collected at the first encounter with the patient, the last measurements will be collected 15 minutes after the intervention in patients who underwent intervention and 1 hour after the first measurement in the control group.
  The temperature of the patients will be measured on the patient's forehead using a digital thermometer. Fever degree will be presented in centigrade (°C).
Blood pressure | The first measurement will be collected at the first encounter with the patient, the last measurements will be collected 15 minutes after the intervention in patients who underwent intervention and 1 hour after the first measurement in the control group.
  Patients' blood pressure will be measured in mmHg using a portable bedside monitor.
Heart rate | The first measurement will be collected at the first encounter with the patient, the last measurements will be collected 15 minutes after the intervention in patients who underwent intervention and 1 hour after the first measurement in the control group.
  Patients' pulses will be measured in beats/minute using a portable bedside monitor.
Saturation | The first measurement will be collected at the first encounter with the patient, the last measurements will be collected 15 minutes after the intervention in patients who underwent intervention and 1 hour after the first measurement in the control group.
  Saturation of patients will be measured in % using a portable bedside monitor
Respiratory rate | The first measurement will be collected at the first encounter with the patient, the last measurements will be collected 15 minutes after the intervention in patients who underwent intervention and 1 hour after the first measurement in the control group.
  The respiratory rate of the patients will be measured by monitoring the patient's chest movements in one minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Isparta Şehir Hastanesi, Isparta, Turkey (Türkiye)